CLINICAL TRIAL: NCT01005537
Title: Single Patient Study to Evaluate Cellular Adoptive Immunotherapy Using Autologous Lymphocytes Following Cyclophosphamide Conditioning for a Single Patient With Metastatic Melanoma
Brief Title: Cyclophosphamide, Autologous Lymphocytes, and Aldesleukin in Treating Patients With Metastatic Melanoma
Status: No longer available | Type: Expanded Access
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Cassian Yee, Fred Hutchinson Cancer Research Center
Other Study IDs: 2355.00; P30CA015704 (NIH); FHCRC-2355.00; IR-6984; CDR0000648071 (Registry Identifier: PDQ)
Record Dates: First submitted 2009-10-30; First posted 2009-11-02 (Estimated); Last update posted 2010-08-06 (Estimated); Status verified 2010-08

CONDITIONS: Melanoma (Skin)
Keywords: stage IV melanoma
MeSH Terms: conditions — Melanoma | interventions — aldesleukin; Cyclophosphamide

INTERVENTIONS:
Biological: aldesleukin — Given IV and orally
Biological: therapeutic autologous lymphocytes — Given IV
Drug: cyclophosphamide — Given IV

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as cyclophosphamide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Biological therapy, such as cellular adoptive immunotherapy using autologous lymphocytes, may stimulate the immune system in different ways and stop tumor cells from growing. Aldesleukin may stimulate the lymphocytes to kill tumor cells. Giving cyclophosphamide together with autologous lymphocytes and aldesleukin may be an effective treatment for metastatic melanoma.

PURPOSE: This phase I/II trial is studying the side effects of giving cyclophosphamide together with autologous lymphocytes and aldesleukin and to see how well it works in treating patients with metastatic melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Assess the safety and toxicity of cellular adoptive immunotherapy with autologous tumor-infiltrating lymphocytes (TIL) following cyclophosphamide conditioning and post-infusion aldesleukin (IL-2) in patients with metastatic melanoma.
* Assess the duration of in vivo persistence of adoptively transferred lymphocytes.

Secondary

* Evaluate the antitumor effect of adoptively transferred autologous TIL following cyclophosphamide conditioning and post-infusion IL-2 in these patients.

OUTLINE: Patients receive cyclophosphamide IV on days -3 and -2 and autologous tumor-infiltrating lymphocytes (TIL) IV on day 0. Beginning 6 hours after TIL infusion, patients receive high-dose aldesleukin (IL-2) IV three times daily on days 0-5 (for up to 14 doses) OR low-dose IL-2 subcutaneously twice daily on days 0-14 (for up to 28 doses). Patients may then receive two additional courses of TILs and low-dose IL-2 (with or without cyclophosphamide), if indicated.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria

* Histopathological documentation of melanoma concurrent with the diagnosis of metastatic disease.
* 18 to 75 years of age and able to tolerate high-dose cyclophosphamide
* Bi-dimensionally measurable disease by palpation on clinical exam, or radiographic imaging (X-ray, CT scan).
* For patients receiving HD-IL-2, normal cardiac stress test within 182 days prior to enrollment is required of all patients over 50 years old or those with an abnormal ECG, any history of cardiac disease, a family history of cardiac disease, hypercholesterolemia or hypertension.
* For leukapheresis, patients must meet the following criteria (any exceptions to this will require prior approval by the Apheresis director and Principal Investigator):

  * Pulse: >45 or < 120
  * Weight: >45 kg
  * Temperature: <38C (<100.4 F)
  * WBC: >3,000
  * HCT: >30%
  * Platelets: >100,000
* ADDITIONAL INCLUSION CRITERIA FOR T CELL INFUSION

Exclusion Criteria

* Significant cardiovascular abnormalities as defined by any one of the following:

  * congestive heart failure,
  * clinically significant hypotension,
  * symptoms of coronary artery disease,
  * presence of cardiac arrhythmias on EKG requiring drug therapy
  * ejection fraction < 50 % (echocardiogram or MUGA)
* Patients with active infections or oral temperature > 38.2 C within 72 hours of study entry or systemic infection requiring chronic maintenance or suppressive therapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2009-06; Primary Completion 2010-10 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Cassian Yee, MD, Principal Investigator — Fred Hutchinson Cancer Center